CLINICAL TRIAL: NCT05721885
Title: A Prospective Single-arm Cohort Study on the Effect of Peri-radiotherapy Nutrition Management on Radiation-induced Oral Mucositis in Patients With Advanced Head and Neck Cancer
Brief Title: Effect of Nutritional Management on RIOM in Patients With Advanced Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jing Yan (Other)
Responsible Party: Sponsor-Investigator, Jing Yan, Chief Physician/Deputy Administrative Director of Oncology Department, Nanjing Drum Tower Hospital, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-496-02
Record Dates: First submitted 2023-01-18; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer; Nutrition Related Cancer; Radiation-Induced Mucositis
Keywords: Head and Neck Cancer; Malnutrition; Radiation-induced Oral Mucositis; nutrition management
MeSH Terms: conditions — Head and Neck Neoplasms; Malnutrition | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Group A: standard treatment group, standard anti-tumor treatment, clinicians in accordance with the NCCN anti-tumor treatment guidelines.
  Group B: peri-radiotherapy nutrition management group, standard anti-tumor therapy combined with peri-radiotherapy nutrition management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peri-radiotherapy nutrition management group (Other): Nutritional management was performed by clinical pharmacists and registered dietitians to develop nutritional intervention strategies based on patient clinical assessment and nutritional assessment. PG-SGA score was 0-3 points, and diet guidance was given. PG-SGA score > 4 points, artificial nutrition intervention was carried out, and the way and amount of nutritional intervention were clarified to achieve the final daily energy and protein target requirements. Nutritional interventions and assessments were adjusted over time.
  Interventions: Behavioral: nutrition management

INTERVENTIONS:
Behavioral: nutrition management — Nutritional management was performed by clinical pharmacists and registered dietitians to develop nutritional intervention strategies based on patient clinical assessment and nutritional assessment. PG-SGA score was 0-3 points, and diet guidance was given. PG-SGA score > 4 points, artificial nutrition intervention was carried out, and the way and amount of nutritional intervention were clarified to achieve the final daily energy and protein target requirements. Nutritional interventions and assessments were adjusted over time.

SUMMARY:
The goal of this clinical trial is to learn about the effect of nutritional management on radiation-induced oral mucositis in patients with advanced head and neck cancer during the peri-radiotherapy period . The main questions it aims to answer are:

* [question 1]Whether whole-course nutritional intervention can improve radiation-induced oral mucositis in patients with HNC.
* [question 2]Whether whole-course nutritional intervention can improve nutritional status and inflammation.

Participants will be treated according to the NCCN guidelines. In addition, clinical pharmacists and registered dietitians provided nutritional intervention strategies based on clinical and nutritional assessments for the patients in the peri-radiotherapy nutrition group.

Researchers will compare clinical routine examination and nutritional indicators between the standard treatment group and the peri-radiotherapy nutrition management group to see if nutrition management effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years old
* Advanced head and neck cancer (III-IV inoperable) is clearly diagnosed
* Predicted survival time > 3 months
* Radical radiotherapy combined with chemotherapy or immunotherapy was performed in our hospital
* The patient has clear consciousness and no communication disorder
* Informed consent and voluntary participation in this study

Exclusion Criteria:

* Patients with previous surgery or radiotherapy for head and neck cancer
* Patients with concurrent or previous history of other tumors
* Distant metastasis
* Patients with allergy, intolerance or contraindication to enteral nutrition or parenteral nutrition
* Severe renal insufficiency (eGFR<30ml/min/1.73m2)
* Combined with poorly controlled metabolic diseases such as diabetes
* Doctors or researchers deem that they are not suitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of radiation-induced oral mucositis (RTOG criteria) | six months
  The Radiation Oncology Group (RTOG) grade of acute radiation injury was used for evaluation, which was divided into 0 to Ⅳ grades. The mild grade included 0, Ⅰ, and Ⅱgrades (grade 0 was no mucosal response; GradeⅠ: erythema, mild pain; GradeⅡ: spotty mucositis with serous exudation), severe grade Ⅲ- IV (Ⅲ: patchy fibrous mucositis with severe pain; Grade IV: necrosis, ulcer, hemorrhage).